CLINICAL TRIAL: NCT05470985
Title: A Phase 2/3, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Oral Ozanimod (RPC1063) in Pediatric Participants With Moderately to Severely Active Crohn's Disease With an Inadequate Response to Conventional Therapy
Brief Title: A Study to Evaluate the Efficacy, Safety, and Drug Levels of Oral Ozanimod in Pediatric Participants With Moderately to Severely Active Crohn's Disease With an Inadequate Response to Conventional Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to business reasons.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM047-023; 2021-005019-30 (EudraCT Number)
Record Dates: First submitted 2022-07-12; First posted 2022-07-22 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ozanimod Dose Level 1 (Experimental)
  Interventions: Drug: Ozanimod
- Ozanimod Dose Level 2 (Experimental)
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Specific dose on specific days
  Other Names: BMS-986374; RPC1063

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, drug levels, and drug effects of ozanimod in pediatric participants with moderately to severely active Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a Pediatric Crohn's Disease Activity Index (PCDAI) score ≥ 30 and a Simple Endoscopic Score for Crohn's Disease (SES-CD) score ≥ 6 (or SES-CD ≥ 4 in participants with isolated ileal disease)
* Participant has an inadequate response, intolerance, or loss of response to at least 1 of the following treatments for Crohn's Disease (CD):

  i) corticosteroids ii) immunomodulators iii) biologic therapy iv) other systemic immunomodulatory therapies for CD

Exclusion Criteria:

* Participant is likely to require, in the physician's judgment, bowel resection within 12 weeks of entry into the study
* Participant has current stoma, ileal-anal pouch anastomosis, fistula that is likely to require, in the physician's judgment, surgical or medical intervention within 12 weeks of entry into the study or need for ileostomy or colostomy
* Participant has extensive small bowel resection (> 100 cm) or known diagnosis of short bowel syndrome or participant requires total parenteral nutrition

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (46):
- United States (19):
  - Local Institution - 0010, Garden Grove, California
  - Local Institution - 0028, Los Angeles, California
  - Local Institution - 0002, Sacramento, California
  - Local Institution - 0009, San Francisco, California
  - Local Institution - 0011, Hartford, Connecticut
  - Local Institution - 0044, Orlando, Florida
  - Local Institution - 0037, Orlando, Florida
  - Local Institution - 0053, Atlanta, Georgia
  - Local Institution - 0059, Indianapolis, Indiana
  - Local Institution - 0038, Springfield, Massachusetts
  - Local Institution - 0006, Detroit, Michigan
  - Local Institution - 0003, Rochester, Minnesota
  - Local Institution - 0016, St Louis, Missouri
  - Local Institution - 0071, Lebanon, New Hampshire
  - Local Institution - 0060, New York, New York
  - Local Institution - 0075, Fort Worth, Texas
  - Local Institution - 0070, Houston, Texas
  - Local Institution - 0008, Seattle, Washington
  - Local Institution - 0040, Tacoma, Washington
- Local Institution - 0045, Joonladup, Western Australia, Australia
- Belgium (6):
  - Local Institution - 0058, Brussels, BRU
  - Local Institution - 0023, Leuven, VBR
  - Local Institution - 0048, Liège, WLG
  - Local Institution - 0062, Liège, WLG
  - Local Institution - 0047, Brussels
  - Local Institution - 0055, Brussels
- Canada (3):
  - Local Institution - 0014, Halifax, Nova Scotia
  - Local Institution - 0001, London, Ontario
  - Local Institution - 0054, Montreal, Quebec
- France (4):
  - Local Institution - 0066, Bron
  - Local Institution - 0065, Caen
  - Local Institution - 0072, Paris
  - Local Institution - 0063, Toulouse
- Germany (2):
  - Local Institution - 0057, Dresden, Saxony
  - Local Institution - 0067, Leipzig, Saxony
- Hungary (2):
  - Local Institution - 0015, Miskolc
  - Local Institution - 0026, Szeged
- Poland (5):
  - Local Institution - 0007, Warsaw, Masovian Voivodeship
  - Local Institution - 0052, Rzeszów, Podkarpackie Voivodeship
  - Local Institution - 0061, Lodz
  - Local Institution - 0031, Warsaw
  - Local Institution - 0033, Warsaw
- Spain (4):
  - Local Institution - 0025, Barcelona, B
  - Local Institution - 0030, Badalona
  - Local Institution - 0035, Barcelona
  - Local Institution - 0017, Madrid

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozanimod 0.46 mg: Participants with moderately to severely active Crohn's Disease with an inadequate response to conventional therapy were administered with 0.46 mg of Ozanimod capsule orally.
- Ozanimod 0.92 mg: Participants with moderately to severely active Crohn's Disease with an inadequate response to conventional therapy were administered with 0.92 mg of Ozanimod capsule orally.
Period: Double Blind Treatment Period
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Started | 3 | 2
Completed | 2 | 1
Not Completed | 1 | 1
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Long Term Extension
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Study terminated by sponsor | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Pediatric Crohn's Disease Activity Index (PCDAI) Score < 10 at Week 64
Description: The PCDAI is an instrument that was developed and validated for numerical assessment of disease activity in children and adolescents with CD. The PCDAI consists of the following 11 variables: Abdominal pain, stools per day, wellbeing, weight, height velocity, abdominal tenderness, peri-rectal disease, extra-intestinal manifestation, hematocrit, erythrocyte sedimentation rate and albumin. The category of severity for each index item is assigned a score: 0=normal;5=mild abnormality; 10= severe abnormality. For hematocrit and erythrocyte SR, the maximum score =5. For albumin level, the maximum score = 10. The PCDAI score is average of 11 variables scoring range of 0 to 100. Mild disease corresponds to scores of 11 to 30; moderate to severe disease corresponds to scores > 30. Remission (no disease activity) is defined as a PCDAI score < 10.
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percentage of Participants Achieving Simple Endoscopic Score for Crohn's Disease (SES-CD) ≤ 2 or SES-CD ≤ 4 Points With no SES-CD Subscore > 1 Point at Week 64
Description: SES-CD assesses the degree of inflammation on the basis of 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these 4 components are assessed in the five segments of the ileum and colon: ileum, right colon, transverse colon, left (descending and sigmoid) colon, and rectum, and is scored on a scale of severity 0 (Normal) to 3 (High). Sub-scores for each segment will be derived by adding component scores within segments. Total SES-CD score is the sum of the sub-scores across the five segments. The sum of each component across all segments ranges from 0 to 15, except for the presence of narrowing where it varies from 0 to 11. The range of the overall SES-CD score is 0-56, with larger scores indicating greater severity of disease.
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Achieve Pediatric Crohn's Disease Activity Index (PCDAI) < 10 at Week 12 Based on Data as Observed
Description: as for outcome 1
Time Frame: Week 12
Population: The Intent to Treat population consist of all randomized participants that receive at least 1 dose of investigational drug. Participants who completed Week 12 visit were only included in the analysis. No participants in Ozanimod 0.46 mg arm completed Week 12 visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Ozanimod 0.92 mg
Number analyzed (Participants) | 1
Percentage of participants | 0

4. Secondary Outcome: Percentage of Participants Who Achieve Simple Endoscopic Score for Crohn's Disease (SES-CD) Decrease From Baseline of ≥ 50% (ER-50) at Week 64
Description: as for outcome 2
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Achieve Simple Endoscopic Score for Crohn's Disease (SES-CD) Decrease From Baseline of ≥ 50% (ER-50) at Week 12 Based on Data as Observed
Description: as for outcome 2
Time Frame: Week 12
Population: The Intent to Treat population consist of all randomized participants that receive at least 1 dose of investigational drug. Only participants who completed week 12 visit are included in the analysis. No participants in Ozanimod 0.46 mg arm completed Week 12 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg
Number analyzed (Participants) | 1
percentage of participants | 0

6. Secondary Outcome: Percentage of Participants Who Achieve Reduction in Pediatric Crohn's Disease Activity Index (PCDAI) Score ≥ 12.5 and a Total PCDAI Score of < 30 Points at Week 64
Description: as for outcome 1
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Achieve Reduction in Pediatric Crohn's Disease Activity Index (PCDAI) Score ≥ 12.5 and a Total PCDAI Score of < 30 Points at Week 12 Based on Data as Observed
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg
Number analyzed (Participants) | 1
percentage of participants | 0

8. Secondary Outcome: Percentage of Adolescents Who Achieve an Average Daily Abdominal Pain Score ≤ 1 Point and an Average Daily Stool Frequency ≤ 3 Points With Abdominal Pain and Stool Frequency no Worse Than Baseline at Week 12 Based on Data as Observed
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as average daily abdominal pain score ≤1 point, and average daily stool frequency ≤ 3 times with AP and SF no worse than baseline at Week 12. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. The AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Ozanimod 0.92mg: Participants with moderately to severely active Crohn's Disease with an inadequate response to conventional therapy were administered with 0.92 mg of Ozanimod capsule orally.
Arm/Group | Ozanimod 0.92mg
Number analyzed (Participants) | 1
percentage of participants | 0

9. Secondary Outcome: Percentage of Adolescents Who Achieve an Average Daily Abdominal Pain Score ≤ 1 Point and an Average Daily Stool Frequency ≤ 3 Points With Abdominal Pain and Stool Frequency no Worse Than Baseline at Week 64
Description: as for outcome 8
Time Frame: Week 64
Population: Data was not collected as no participants in the study completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Stool Frequency (SF) Score at Week 64
Description: SF was defined number of liquid or soft stools per day.
Time Frame: Baseline and Week 64
Population: Data was not collected as no participants completed Week 64 visit. Pre-specified to assess change at Week 64.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Abdominal Pain (AP) Score at Week 64
Description: Participants entered Reponses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score. The AP score was graded on severity of 0 (none) to 3 (severe) scale.
Time Frame: Baseline and Week 64
Population: Data was not collected as no participants completed Week 64 visit. Pre-specified to assess change at Week 64.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Adolescents Who Achieve Crohn's Disease Activity Index (CDAI) Score < 150 at Week 12 Based on Data as Observed
Description: The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease (CD). The CDAI uses a questionnaire with 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. The sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: Week 12
Population: The Intent to Treat population consist of all randomized participants that receive at least 1 dose of investigational drug. Participants who completed week 12 visit were included in the analysis. No participants in Ozanimod 0.46 mg arm completed Week 12 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92mg
Number analyzed (Participants) | 1
percentage of participants | 0

13. Secondary Outcome: Percentage of Adolescents Who Achieve Crohn's Disease Activity Index (CDAI) Score < 150 at Week 64
Description: as for outcome 12
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Adolescents Who Achieve Crohn's Disease Activity Index (CDAI) Reduction From Baseline of ≥ 100 Points or CDAI Score < 150 at Week 64
Description: as for outcome 12
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Adolescents Who Achieve Crohn's Disease Activity Index (CDAI) Reduction From Baseline of ≥ 100 Points or CDAI Score < 150 at Week 12 Based on Data as Observed
Description: as for outcome 12
Time Frame: Week 12
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92mg
Number analyzed (Participants) | 1
percentage of participants | 0

16. Secondary Outcome: Percentage of Participants Who Achieve a Pediatric Crohn's Disease Activity Index (PCDAI) Score < 10 at Week 64 While Remaining Corticosteroid Free in the Prior 12 Weeks
Description: as for outcome 1
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Percentage of Adolescents Who Achieve a Pediatric Crohn's Disease Activity Index (PCDAI) Score < 10 at Week 64 While Remaining Corticosteroid Free in the Prior 12 Weeks
Description: as for outcome 1
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percentage of Participants Who Achieve a Crohn's Disease Activity Index (CDAI) Score < 150 at Week 64 While Remaining Corticosteroid Free in the Prior 12 Weeks
Description: as for outcome 12
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Percentage of Participants Achieving Simple Endoscopic Score for Crohn's Disease (SES-CD) ≤ 2 or SES-CD ≤ 4 Points With no SES-CD Subscore > 1 Point at Week 12 Based on Data as Observed
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92mg
Number analyzed (Participants) | 1
percentage of participants | 0

20. Secondary Outcome: Steady State Systemic Exposures of Ozanimod at Week 20 and Throughout the Study
Description: Blood samples were collected to assess steady state exposure of ozanimod.
Time Frame: Week 20 and up to end of study (Week 64)
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Absolute Lymphocyte Count at Week 12 Based on Data as Observed
Description: Blood samples were collected to assess lymphocyte count.
Time Frame: Baseline (Day 1) and Week 12
Population: The Intent to Treat population consist of all randomized participants that receive at least 1 dose of investigational drug. Participants who completed Week 12 visit were only considered in the analysis. No participants in Ozanimod 0.46 mg arm completed Week 12 visit.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Ozanimod 0.92mg
Number analyzed (Participants) | 1
10^9 cells per liter | 0.66 (NA) — Insufficient number of participants to calculate SD

22. Secondary Outcome: Absolute Lymphocyte Count at Week 64
Description: Blood samples were collected to assess lymphocyte count.
Time Frame: Week 64
Population: Data was not collected as no participants completed Week 64 visit.
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92 mg
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Serious Adverse Events (SAEs) is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization; results significant disability; or is a congenital anomaly/birth defect.
Time Frame: From first dose (Day 1) and up to Week 12
Population: The Intent to Treat population consist of all randomized participants that receive at least 1 dose of investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ozanimod 0.46 mg | Ozanimod 0.92mg
Number analyzed (Participants) | 3 | 2
Participants
  Adverse Events | 3 | 2
  Serious Adverse Events | 0 | 0
  Adverse events leading to Discontinuation | 0 | 0
  Adverse Events of Special Interest | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, serious adverse events and non serious adverse events were collected from Day 1 to Week 12.
Description: The Intent to Treat population consist of all randomized participants that receive at least 1 dose of investigational drug.
Groups:
- Ozanimod 0.46mg: Participants with moderately to severely active Crohn's Disease with an inadequate response to conventional therapy were administered with 0.46 mg of Ozanimod capsule orally.
Arm/Group | Ozanimod 0.46mg | Ozanimod 0.92mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod 0.46mg (N=3) | Ozanimod 0.92mg (N=2)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod 0.46mg (N=3) | Ozanimod 0.92mg (N=2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT05470985/Prot_SAP_000.pdf